CLINICAL TRIAL: NCT01377922
Title: A Phase 3, Double-blind, Placebo-controlled, Randomized Discontinuation Study Followed by Open-label Extension Evaluating Efficacy and Safety of Amifampridine Phosphate in Patients With Lambert-Eaton Myasthenic Syndrome (LEMS)
Brief Title: A Phase 3 Study of Amifampridine Phosphate in Patients With Lambert Eaton Myasthenic Syndrome (LEMS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LMS-002
Record Dates: First submitted 2011-06-17; First posted 2011-06-22 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Lambert Eaton Myasthenic Syndrome
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome | interventions — Amifampridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo tablets administered 3-4 times a day (to the individual patient's tablet count of active at baseline) over 2 weeks.
  Interventions: Drug: Placebo
- Amifampridine Phosphate (Experimental): Amifampridine, 30-80 mg given 3-4 times per day with a maximum single dose of 20 mg (2 x 10 mg tablets), for 2 weeks.
  Interventions: Drug: Amifampridine Phosphate

INTERVENTIONS:
Drug: Amifampridine Phosphate — Amifampridine, 30-80 mg given 3-4 times per day with a maximum single dose of 20 mg (2 x 10 mg tablets), for 2 weeks.
  Other Names: 3,4-diaminopyridine phosphate; 3,4-DAP phosphate
  Arms: Amifampridine Phosphate
Drug: Placebo — Matching placebo tablets administered 3-4 times a day (to the individual patient's tablet count of active at baseline) over 2 weeks.
  Arms: Placebo

SUMMARY:
A Phase 3 study to evaluate the efficacy and safety of Amifampridine Phosphate in patients with Lambert-Eaton Myasthenic Syndrome (LEMS).

DETAILED DESCRIPTION:
This multicenter, double-blind, placebo-controlled, randomized (1:1) discontinuation study is a 4-part study designed to evaluate the efficacy and safety of multiple dose administration of amifampridine phosphate in patients with LEMS. Data from parts 2 and 3 (the double-blind parts of the study) are presented in this record.

ELIGIBILITY:
Inclusion Criteria: Individuals eligible to participate in this study must meet all of the following inclusion criteria:

* ≥18 years of age
* Confirmed diagnosis of LEMS
* Normal respiratory function
* Normal swallowing function
* If receiving peripherally acting cholinesterase inhibitors a stable dose is required for at least 7 days prior to Screening.
* If receiving oral immunosuppressants a stable dose is required for at least 90 days prior to Screening.
* Negative pregnancy test for females of childbearing potential
* If sexually active, willing to use 2 acceptable methods of contraception
* Willing to perform all study procedures as physically possible.
* Willing and able to provide written informed consent after the nature of the study has been explained and prior to the start of any research-related procedures.

Exclusion Criteria: Individuals who meet any of the following exclusion criteria are not eligible to participate in the study:

* History of epilepsy or seizure.
* Known active brain metastasis.
* Use of Fampridine (4-aminopyridine), and any form of 3,4-diaminopyridine other than the IP provided, such as amifampridine base or Firdapse, during the study.
* Use of medications known to lower the epileptic threshold within 7 days or 5 half-lives.
* Use of medications which inhibit neuromuscular junction function within 7 days or 5 half-lives.
* Use of IVIG, plasmapheresis (plasma exchange), or immunoadsorption within 90 days
* Use of guanidine hydrochloride within 7 days
* Use of rituximab within 12 months
* History of drug allergy to any pyridine-containing substances or any amifampridine phosphate excipient(s).
* Use of any other investigational productwithin 30 days
* Treatment with a concomitant medication that prolongs the QT/QTc interval within 7 days or 5 half-lives.
* Treatment with sultopride (4-amino-N-[(1-ethylpyrrolidin-2-yl)methyl]-5-ethylsulfonyl-2-methoxybenzamide) within 7 days.
* An abnormal electrocardiogram (ECG).
* Documented history of arrhythmias.
* History of additional risk factors for torsade de pointes.
* Breastfeeding or pregnant or planning to become pregnant (self or partner) at any time during the study.
* Likely or expected to require treatment for cancer within 3 months (90 days) after entering.
* History of severe renal impairment or evidence of severe renal impairment
* Any condition that places the patient at high risk of poor treatment compliance or of not completing the study.
* History of uncontrolled asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Gorodetzky, MD, PhD, Study Director — Chief Medical Officer
Locations (14):
- United States (6):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Los Angeles, California
  - Palo Alto, California
  - Kansas City, Kansas
  - New York, New York
- Lyon, France
- Germany (2):
  - Munich, Bavaria
  - Berlin
- Pécs, Hungary
- Warsaw, Poland
- Moscow, Russia
- Belgrade, Serbia
- Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 clinical sites in 8 countries, including France, Germany, Hungary, Poland, Russia, Serbia, Spain, and the United States.
  The study was conducted from 03Jun2011 to 08Jul2016.
Pre-assignment Details: Open-label Run-in (Part 1): titration to the optimal amifampridine dose (well tolerated and resulted in a ≥3 point improvement in QMG score from Screening for patients without previous amifampridine use) for each individual patient. Patients who did not receive amifampridine prior to Run-in and who did not reach the optimal dose were discontinued.
Groups:
- Part 2 and Part 3 Placebo: Matching placebo tablets, administered 3-4 times a day for 2 weeks.
  Placebo tablets indistinguishable from amifampridine phosphate tablets. The placebo was administered consistent with the dose and dose regimen of amifampridine phosphate.
- Part 2 and Part 3 Amifampridine Phosphate: Matching amifampridine phosphate tablets, 10 mg, administered 3-4 times a day for 2 weeks.
  Amifampridine Phosphate: 30-80 mg given 3-4 times per day with a maximum single dose of 20 mg (2 x 10 mg tablets).
Period: Overall Study
Arm/Group | Part 2 and Part 3 Placebo | Part 2 and Part 3 Amifampridine Phosphate
Started | 22 | 16
Completed | 21 | 16
Not Completed | 1 | 0
Not completed — rescue tx after part 2, entered part 4 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 2 and Part 3 Placebo | Part 2 and Part 3 Amifampridine Phosphate | Total
Number analyzed (Participants) | 22 | 16 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (17.57) | 51.6 (12.05) | 51.5 (15.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 22 | 12 | 34
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 13 | 34
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 1 | 2
Was the patient taking amifampridine (base or phosphate) immediately prior to enrollment? [Count of Participants; unit: Participants]
  Yes | 7 | 3 | 10
  No | 15 | 13 | 28
If yes, number of continuous days of amifampridine exposure immediately prior to enrollment [Mean (Standard Deviation); unit: days] — Population: Data only for those subjects (7 in the placebo group, 3 in the amifampridine group) who were taking amifampridine prior to enrollment.
  days
    number analyzed (Participants) | 7 | 3 | 10
    (all) | 1287.1 (1525.73) | 2143.3 (3080.16) | 1544.0 (1957.36)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Quantitative Myasthenia Gravis (QMG) at 14 Days
Description: The QMG is a physician-rated test including 13 assessments, including facial strength, swallowing, grip strength, and duration of time that limbs can be maintained in outstretched positions. Each of the 13 items is scored from 0 (none) to 3 (severe). The total score can range from 0 to 39. Increased QMG total score correlates to worsening symptoms of LEMS.
Time Frame: Assessment at Baseline and Day 14
Measure: Mean (Standard Deviation); unit: QMG Score
Groups:
- Placebo: Matching placebo tablets administered 3-4 times a day over 2 weeks.
  Placebo: Matching number of tablets to the individual patient's tablet count of active at baseline.
- Amifampridine Phosphate: Matching amifampridine phosphate tablets, 10 mg, administered 3-4 times a day for 2 weeks.
  Amifampridine Phosphate: 30-80 mg given 3-4 times per day with a maximum single dose of 20 mg (2 x 10 mg tablets).
Arm/Group | Placebo | Amifampridine Phosphate
Number analyzed (Participants) | 21 | 16
QMG Score
  Baseline | 5.6 (3.99) | 6.4 (3.22)
  Day 14 | 7.9 (2.85) | 6.7 (4.09)
  Change from Baseline | 2.2 (2.93) | 0.3 (2.60)
Statistical Analysis 1: Comparison: Placebo vs Amifampridine Phosphate; Test type: Other — Estimated via a MMRM with change from baseline (Day 1, Part 2), Day 8, and Day 14 as the dependent variable and terms for treatment, time (Day 8, Day 14), treatment-by-time interaction, and double-blind baseline QMG score as fixed effects and patient as a random effect. The model assumed time effect to be random between patients; p = 0.0452, Mixed Models Analysis; Pairwise contrast at Day 14 from MMRM model

2. Primary Outcome: Change in SGI Score
Description: Subject Global Impression (SGI) is a measure of changes in subject's perception of change in overall wellbeing.
  The patient is asked to use the 7-point scale below to rate their impression of the effects of the study medication during the preceding 3 days on their physical well being.
  1. Terrible
  2. Mostly dissatisfied
  3. Mixed
  4. Partially satisfied
  5. Mostly satisfied
  6. Pleased
  7. Delighted
Time Frame: Assessment at Baseline and Day 14
Population: FAS
Measure: Mean (Standard Deviation); unit: SGI score
Arm/Group | Placebo | Amifampridine Phosphate
Number analyzed (Participants) | 21 | 16
SGI score
  Baseline | 5.9 (1.22) | 5.6 (1.26)
  Day 14 | 3.2 (1.7) | 4.9 (1.57)
  Change from Baseline | -2.7 (2.29) | -0.7 (1.82)
Statistical Analysis 1: Comparison: Placebo vs Amifampridine Phosphate; Estimated via a MMRM with change from baseline (Day 1, Part 2), Day 8, and Day 14 as the dependent variable and terms for treatment, time (Day 8, Day 14), treatment-by-time interaction, and double-blind baseline SGI score as fixed effects and patient as a random effect. The model assumed time effect to be random between patients; Test type: Other; p = 0.0028, Mixed Models Analysis — Pairwise contrast at Day 14 from MMRM model

3. Secondary Outcome: Change From Baseline Timed 25 Foot Walking Test (T25FW) at 14 Days
Description: The T25FW test, a component of the Multiple Sclerosis Functional Composite, was a quantitative mobility and leg function performance test based on a timed 25-foot walk (National Multiple Sclerosis Society). The patient was directed to walk a clearly marked 25-foot course as quickly and safely as possible. Following a rest of at least 5 minutes, the timed 25-foot walk was repeated. Patients could use assistive devices, such as canes, crutches, or walkers.
  All data were normalized to the number of feet per minute, so if the patient walked 25 feet in less than a minute, the result was a speed greater than 25 feet/minute.
  The measurement for the T25FW test was the average speed, expressed in feet/minute, of the 2 completed walks.
Time Frame: Assessment at Baseline and Day 14
Measure: Mean (Standard Deviation); unit: feet/minute
Arm/Group | Placebo | Amifampridine Phosphate
Number analyzed (Participants) | 21 | 16
feet/minute
  Baseline | 255 (111) | 254 (126)
  Day 14 | 244 (116) | 253 (126)
  Change from Baseline | -10.4 (53.1) | -1.46 (52.5)
Statistical Analysis 1: Comparison: Placebo vs Amifampridine Phosphate; Estimated via a MMRM with change from baseline (Day 1, Part 2), Day 8, and Day 14 as the dependent variable and terms for treatment, time (Day 8, Day 14), treatment-by-time interaction, and double-blind baseline T25FW walking speed as fixed effects and patient as a random effect. The model assumed time effect to be random between patients; Test type: Other; p = 0.6274, Mixed Models Analysis

4. Secondary Outcome: Change in CGI-I Score
Description: The Investigator completed the 7-point CGI I, based on changes in symptoms, behavior, and functional abilities, at the protocol-specified time points compared to the patient's condition at Day 0.
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: CGI-I score
Arm/Group | Placebo | Amifampridine Phosphate
Number analyzed (Participants) | 21 | 16
CGI-I score
  Baseline | 2.5 (0.98) | 2.6 (0.63)
  Day 14 | 4.8 (1.45) | 3.6 (1.50)
Statistical Analysis 1: Comparison: Placebo vs Amifampridine Phosphate; Estimated via a MMRM with change from baseline (Day 1, Part 2), Day 8, and Day 14 as the dependent variable and terms for treatment, time (Day 8, Day 14), treatment-by-time interaction as fixed effects and patient as a random effect. The model assumed time effect to be random between patients; Test type: Other; p = 0.0267, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: The reporting period for non-serious AEs was the first administration of study drug through the termination visit or at the early termination visit. The reporting period for SAEs began after a signed ICF was obtained and continued through 4 weeks after the last dose or at the early termination visit.
Description: For this study, the following additional events were considered SAEs:
  * A generalized tonic-clonic convulsion/seizure;
  * A normal liver function test for a patient at Screening, but the patient developed the following constellation of findings:
    * ALT or AST >3 times the ULN;
    * total bilirubin >2 times the ULN; and
    * no other explanation, such as concurrent liver disease or treatment with a potentially hepatotoxic concurrent medication, was found.
Arm/Group | Part 2 and Part 3 Placebo | Part 2 and Part 3 Amifampridine Phosphate
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/16
Other Adverse Events (participants affected / at risk) | 6/21 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 2 and Part 3 Placebo (N=21) | Part 2 and Part 3 Amifampridine Phosphate (N=16)
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0
Pulpitis dental (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Asthenia (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less